CLINICAL TRIAL: NCT00013533
Title: Pilot Study of Non-Myeloablative, HLA-Matched Allogeneic Stem Cell Transplantation for Pediatric Hematopoietic Malignancies
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010125; 01-C-0125; NCT00020592 (obsolete NCT alias)
Record Dates: First submitted 2001-03-20; First posted 2001-03-21 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2015-05-07

CONDITIONS: Hodgkin Lymphoma; Lymphocytic Leukemia; Mixed Cell Leukemia; Myelodysplastic Syndrome; Non Hodgkin's Lymphoma; CML; ALL; AML; Lymphoma
Keywords: Leukemia; Myelodysplastic Syndrome; Bone Marrow Transplant; Pediatric Oncology; Lymphoma; Efficacy; Safety; Childhood Cancer
MeSH Terms: conditions — Hodgkin Disease; Leukemia, Lymphoid; Leukemia, Biphenotypic, Acute; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Lymphoma; Leukemia; Neoplasms | interventions — Stem Cell Transplantation

ARMS (1):
- 1 (Experimental): Transplant with Induction Therapy
  Interventions: Procedure: Stem cell transplantation

INTERVENTIONS:
Procedure: Stem cell transplantation — >3 x 106/kg CD34+ stem cells by IV infusion

SUMMARY:
Background:

* Allogeneic blood and marrow stem cell transplantation (BMT) plays an important role in the curative treatment of a number of pediatric malignancies. Unfortunately, the success of conventional allogeneic BMT is limited in part by the multiple toxicities associated with myeloablative preparative regimens.
* Non-myeloablative pre-transplant regimens are associated with less toxic side effects than standard BMT. Recently, a novel immunosuppressive, non-myeloablative pre-transplant chemotherapy regimen has been shown to facilitate complete donor engraftment in an adult trial at the NCI.

Objectives:

The primary objective of this protocol is to evaluate the efficacy and safety of this treatment approach in pediatric patients with hematopoietic malignancies

Eligibility:

Inclusion Criteria

Age: Patient must be greater than or equal to 5 years and less than 22 years of age.

Diagnosis:

* Hodgkin s and Non-Hodgkin s Lymphoma: Refractory disease or relapse after salvage regimen.
* Acute Myelogenous Leukemia: History of bone marrow relapse in remission (CR) #2 or greater.
* Acute Lymphocytic Leukemia: History of bone marrow relapse in CR #2 or greater (CR#1 with Philadelphia chromosome positive or prior induction failure).
* Acute Hybrid Leukemia including mixed lineage, biphenotypic and undifferentiated: History of bone marrow relapse in CR #2 or greater (CR#1 with Philadelphia chromosome positive or prior induction failure).
* Myelodysplastic Syndrome: RAEB or RAEB-t with less than 10% blasts in marrow and blood.
* Chronic Myelogenous Leukemia: Chronic phase or accelerated phase with less than 10% blasts in marrow and blood.
* Juvenile Myelomonocytic Leukemia: less than 10% blasts in marrow and blood.

Prior Therapy: Chemotherapy to achieve above criteria allowed. Prior BMT allowed as long as at least day 100+ post-prior BMT, no evidence of GVHD, and no detectable residual donor chimerism.

Donor: First degree related donors, who are HLA matched (single HLA-A or B locus mismatch allowed), weight greater than or equal to 15 kilograms, and who meet standard donation criteria will be considered. The same donor from a prior BMT is allowed.

ECOG Performance Status: 0, 1, or 2. and life expectancy: greater than 3 months.

Liver Function: Serum direct bilirubin less than 2.0 mg/dL and serum ALT and AST values less than or equal to 2.5x upper limit of normal. (Values above these levels may be accepted if due to malignancy.)

Renal Function: Age adjusted normal serum creatinine or Cr clearance greater than or equal to 60 mL/min/1.73 m(2).

Pulmonary Function: DLCO greater than or equal to 50%.

Cardiac Function: LVEF greater than or equal to 45% by MUGA or LVSF greater than or equal to 28% by ECHO

Exclusion Criteria

* Active CNS malignancy: Tumor mass on CT or leptomeningeal disease. (Patients with a history of CNS involvement and no current evidence of CNS disease are allowed.)
* HIV infection, active hepatitis B or C infection: HbSAg or HCV seropositive and elevated liver transaminases.
* Fanconi Anemia.
* Lactating or pregnant females.

Design:

Pilot Study

* Initial evaluation: Patient and donor will be screened for eligibility. G-CSF primed bone marrow derived stem cells will be collected from the donor.
* Induction/Consolidation chemotherapy: 1 to 3 cycles will be given every 22 days depending on disease response, CD4 count, and toxicities.
* Lymphoma: fludarabine, etoposide, doxorubicin, vincristine, cyclophohamide, prednisone, and filgrastim (EPOCH-fludarabine).
* Leukemia and MDS: Fludarabine, cytarabine, and filgrastim (FLAG).
* Transplantation: Fludarabine and cyclophosphamide will be administered over 4 days followed by bone marrow transplant. Patients will remain hospitalized until bone marrow recovery. Patients will be monitored closely at the NIH for at least 100 days post-BMT.
* Post-transplant CNS prophylaxis for ALL: Standard post-transplant CNS prophylaxis will be employed with intrathecal methotrexate to decrease the risk of CNS relapse for all patients with ALL.
* Total number of recipient and donors to be accrued is 56.

DETAILED DESCRIPTION:
Background:

* Allogeneic blood and marrow stem cell transplantation (BMT) plays an important role in the curative treatment of a number of pediatric malignancies. Unfortunately, the success of conventional allogeneic BMT is limited in part by the multiple toxicities associated with myeloablative preparative regimens.
* Non-myeloablative pre-transplant regimens are associated with less toxic side effects than standard BMT. Recently, a novel immunosuppressive, non-myeloablative pre-transplant chemotherapy regimen has been shown to facilitate complete donor engraftment in an adult trial at the NCI.

Objectives:

The primary objective of this protocol is to evaluate the efficacy and safety of this treatment approach in pediatric patients with hematopoietic malignancies

Eligibility:

Inclusion Criteria

Age: Patient must be greater than or equal to 5 years and less than 22 years of age.

Diagnosis:

* Hodgkin s and Non-Hodgkin s Lymphoma: Refractory disease or relapse after salvage regimen.
* Acute Myelogenous Leukemia: History of bone marrow relapse in remission (CR) #2 or greater.
* Acute Lymphocytic Leukemia: History of bone marrow relapse in CR #2 or greater (CR#1 with Philadelphia chromosome positive or prior induction failure).
* Acute Hybrid Leukemia including mixed lineage, biphenotypic and undifferentiated: History of bone marrow relapse in CR #2 or greater (CR#1 with Philadelphia chromosome positive or prior induction failure).
* Myelodysplastic Syndrome: RAEB or RAEB-t with less than 10% blasts in marrow and blood.
* Chronic Myelogenous Leukemia: Chronic phase or accelerated phase with less than 10% blasts in marrow and blood.
* Juvenile Myelomonocytic Leukemia: less than 10% blasts in marrow and blood.

Prior Therapy: Chemotherapy to achieve above criteria allowed. Prior BMT allowed as long as at least day 100+ post-prior BMT, no evidence of GVHD, and no detectable residual donor chimerism.

Donor: First degree related donors, who are HLA matched (single HLA-A or B locus mismatch allowed), weight greater than or equal to 15 kilograms, and who meet standard donation criteria will be considered. The same donor from a prior BMT is allowed.

ECOG Performance Status: 0, 1, or 2. and life expectancy: greater than 3 months.

Liver Function: Serum direct bilirubin less than 2.0 mg/dL and serum ALT and AST values less than or equal to 2.5x upper limit of normal. (Values above these levels may be accepted if due to malignancy.)

Renal Function: Age adjusted normal serum creatinine or Cr clearance greater than or equal to 60 mL/min/1.73 m(2).

Pulmonary Function: DLCO greater than or equal to 50%.

Cardiac Function: LVEF greater than or equal to 45% by MUGA or LVSF greater than or equal to 28% by ECHO

Exclusion Criteria

* Active CNS malignancy: Tumor mass on CT or leptomeningeal disease. (Patients with a history of CNS involvement and no current evidence of CNS disease are allowed.)
* HIV infection, active hepatitis B or C infection: HbSAg or HCV seropositive and elevated liver transaminases.
* Fanconi Anemia.
* Lactating or pregnant females.

Design:

Pilot Study

* Initial evaluation: Patient and donor will be screened for eligibility. G-CSF primed bone marrow derived stem cells will be collected from the donor.
* Induction/Consolidation chemotherapy: 1 to 3 cycles will be given every 22 days depending on disease response, CD4 count, and toxicities.
* Lymphoma: fludarabine, etoposide, doxorubicin, vincristine, cyclophohamide, prednisone, and filgrastim (EPOCH-fludarabine).
* Leukemia and MDS: Fludarabine, cytarabine, and filgrastim (FLAG).
* Transplantation: Fludarabine and cyclophosphamide will be administered over 4 days followed by bone marrow transplant. Patients will remain hospitalized until bone marrow recovery. Patients will be monitored closely at the NIH for at least 100 days post-BMT.
* Post-transplant CNS prophylaxis for ALL: Standard post-transplant CNS prophylaxis will be employed with intrathecal methotrexate to decrease the risk of CNS relapse for all patients with ALL.
* Total number of recipient and donors to be accrued is 56.

ELIGIBILITY:
* INCLUSION CRITERIA PATIENTS:

Patients with the following diagnoses will be considered:

* Hodgkin's and Non-Hodgkin's Lymphoma: Refractory (non-CR) to primary treatment regimen; Refractory (non-CR) to or relapse after salvage regimen.
* Acute Myelogenous Leukemia (AML): History of bone marrow relapse it CR number 2 or greater.
* Acute Lymphocytic Leukemia (ALL): History of bone marrow relapse in CR number 2 or greater; complete remission #1 with Philadelphia chromosome positive or prior induction failure (subsequent induction regimen required to achieve CR).
* Acute hybrid leukemia including mixed lineage, biphenotypic, and undifferentiated (AUL): History of bone marrow relapse in CR number 2 or greater; Complete remission #1 with Philadelphia chromosome positive or prior induction failure (second induction regimen required to achieve (CR).
* Myelodysplastic Syndrome (MDS) excluding refractory anemia (RA) and RA with ringed sideroblasts (RARS): blasts less than 10% in marrow and blood.
* Chronic Myelogenous Leukemia (CML): Chronic Phase; Accelerated Phase with blasts less than 10% in marrow and blood.
* Juvenile Myelomonocytic Leukemia (JMML, J-CML): Blasts less than 10% in marrow and blood.

Patients must be greater than or equal to 4 years and less than 22 years of age.

Prior chemotherapy: Chemotherapy to achieve above noted criteria allowed. Prior autologous BMT allowed. Prior allogeneic BMT allowed as long as at least day +100 post-prior BMT, and no evidence of ongoing active GVHD.

Availability of 5 or 6 antigen genotypic HLA-matched first-degree relative donor (single HLA-A or B locus mismatch allowed).

Performance status of 0,1, or 2.

Life expectancy greater than 3 months.

Liver function: serum direct bilirubin less than 2.0 mg/dL, and serum ALT and AST values less than or equal to 2.5 times the upper limit of normal. Values above these levels may be accepted, at the discretion of the PI, if such elevations are thought to be due to malignancy (excluding acute leukemia).

Renal function: age-adjusted normal serum creatinine or a creatinine clearance greater than or equal to 60 mL/min/1.73 m(2).

Pulmonary function: DLCO corrected for hemoglobin and alveolar volume greater than or equal to 50% of predicted.

Left ventricular function: Ejection fraction greater than or equal to 45% by MUGA or shortening fraction greater than or equal to 28% by ECHO.

Ability to give informed consent. For patients less than 18 years old their legal guardian must give informed consent. Pediatric patients will be included in age appropriate discussion in order to obtain verbal assent.

Durable power of attorney form completed (patients greater than 18 years of age only).

Patients must not have an active CNS malignancy as defined by: lymphoma (tumor mass on CT scan or leptomeningeal disease), Leukemia (CNS 2 or CNS 3 classification), or NB (History of CNS involvement with no current evidence of CNS malignancy is NOT an exclusion).

Patients must not be HIV positive.

Patients must not have active hepatitis B or C infection as defined by seropositive for hepatitis B (HbSAg) or hepatitis C and elevated liver transaminases.

Female patients must not be lactating or pregnant (due to risk to fetus or newborn).

Patients must not have high risk of inability to comply with transplant protocol as determined by principal investigator, social work, and BMT team.

Patients must not have Fanconi Anemia (FA): patients with MDS must have a negative FA test.

INCLUSION CRITERIA DONOR:

First degree relative with genotypic identity at 5 or 6 HLA loci (single HLA-A or B locus mismatch allowed).

Weight of greater than or equal to 15 kilograms.

Adequate venous access for peripheral apheresis, or consent to use a temporary central venous catheter for apheresis (on Cohort #2, for possible future cell collection if needed).

Ability to give informed consent. For donors less than 18 years of age, he/she must be the oldest eligible donor, their legal guardian must give informed consent, the donor must give verbal assent, and he/she must be cleared by social work and a mental health specialist to participate.

Donor selection criteria will be in accordance with NIH/CC Department of Transfusion Medicine standards.

EXLCUSION CRITERIA PATIENT:

Active CNS malignancy as defined by:

* Lymphoma: tumor mass on CT scan or leptomeningeal disease
* Leukemia: CNS 2 or CNS 3 classification
* NB: History of CNS involvement with no current evidence of CNS malignancy is NOT an exclusion.

HIV positive.

Active hepatitis B or C infection as defined by seropositive for hepatitis B (HbsAg) or hepatitis C and elevated liver transaminases.

Lactating or pregnant females.

High risk of inability to comply with transplant protocol as determined by principal investigator, social work, and BMT team.

Fanconi Anemia (FA): Patients with MDS must have a negative FA test.

EXCLUSION CRITERIA DONOR:

History of medical illness which in the estimation of the PI or DTM physician poses prohibitive risk to donation including, but not limited to stroke, hypertension that is not controlled by medication, or heart disease. Individuals with symptomatic angina or a history of coronary artery bypass grafting or angioplasty will not be eligible. History of congenital hematologic, immunologic, or metabolic disorder which in the estimation of the PI poses prohibitive risk to the recipient.

Anemia (Hb less than gm/dl) or thrombocytopenia (less than 100,000/ul).

Lactating or pregnant females.

HIV positive.

Seropositive for hepatitis B (HbsAg) or hepatitis C.

High risk of inability to comply with transplant protocol as determined by principal investigator, social work, and BMT team.

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2001-03-14; Primary Completion 2008-03-01 (Actual); Study Completion 2015-05-07 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy and safety of this chemotherapy regimen in facilitating donor engraftment after allogeneic bone marrow transplantation (BMT).
Safety/Efficacy | 5 years

SECONDARY OUTCOMES:
Toxicity of regimen | 5 years
To determine the toxicity of this non-myelablative allogeneic BMT regimen.
fludarabine-based induction reducing T-cells | 5 years
immune suppression | 5 years
IL-7 levels | 5 years
cytokine profiles | 5 years
response rates and DFS | 5 years
incidence and severity of GVHD | 5 years
response rates, DFS rates, and incidence and severity ofGVHD following withdrawal of immunosuppression and donorlymphocyte infusions (DLI) for patients who developprogressive disease after day +28 post-transplant | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Terry J Fry, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kantarjian HM, Deisseroth A, Kurzrock R, Estrov Z, Talpaz M. Chronic myelogenous leukemia: a concise update. Blood. 1993 Aug 1;82(3):691-703. No abstract available. PMID 8338938
- [Background] Pui CH, Evans WE. Acute lymphoblastic leukemia. N Engl J Med. 1998 Aug 27;339(9):605-15. doi: 10.1056/NEJM199808273390907. No abstract available. PMID 9718381
- [Background] Rivera GK, Buchanan G, Boyett JM, Camitta B, Ochs J, Kalwinsky D, Amylon M, Vietti TJ, Crist WM. Intensive retreatment of childhood acute lymphoblastic leukemia in first bone marrow relapse. A Pediatric Oncology Group Study. N Engl J Med. 1986 Jul 31;315(5):273-8. doi: 10.1056/NEJM198607313150501. PMID 3523250